CLINICAL TRIAL: NCT05838768
Title: An Open-label, Multi-center Phase I/Ib Dose Finding and Expansion Study of HRO761 as Single Agent and in Combinations in Patients With Microsatellite Instability-High or Mismatch Repair Deficient Advanced Solid Tumors.
Brief Title: Study of HRO761 Alone or in Combination in Cancer Patients With Specific DNA Alterations Called Microsatellite Instability or Mismatch Repair Deficiency.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHRO761A12101; 2022-502314-93-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: MSIhi or dMMR Advanced Unresectable or Metastatic Solid Tumors, Including Colorectal Cancers
Keywords: Phase I/Ib; MSIhi (Microsatellite Instability-High); dMMR (Mismatch Repair Deficient); solid tumors; CRC (Colorectal cancer); advanced cancer; metastatic; HRO761; pembrolizumab; irinotecan
MeSH Terms: conditions — Turcot syndrome; Colorectal Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Irinotecan

STUDY DESIGN:
Masking Description: This is an open label study. Treatment will be open to patients, Investigator staff, persons performing the assessments and the Sponsor clinical trial team.
  For the dose escalation and dose expansion, no randomization will be performed. For the dose optimization (HRO761 single agent arm only), patients will be equally randomized to the two selected HRO761 single agent treatment dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: HRO761 single agent (Experimental): phase Ib (Dose finding (Escalation and Optimization) and expansion)
  Interventions: Drug: HRO761
- B: HRO761 + pembrolizumab (Experimental): phase Ib (Dose escalation and expansion)
  Interventions: Drug: HRO761; Biological: pembrolizumab
- C: HRO761 + irinotecan (Experimental): phase Ib (Dose escalation and expansion)
  Interventions: Drug: HRO761; Drug: irinotecan

INTERVENTIONS:
Drug: HRO761 — Tablet
Biological: pembrolizumab — Concentrate for solution for infusion
  Arms: B: HRO761 + pembrolizumab
Drug: irinotecan — Concentrate for solution for infusion
  Arms: C: HRO761 + irinotecan

SUMMARY:
The main purpose of the study is to evaluate the safety and tolerability of HRO761 and identify the recommended dose(s), i.e., the optimal safe and active dose of HRO761 alone or in combination with pembrolizumab or irinotecan that can be given to patients who have cancers with specific molecular alterations called MSIhi (Microsatellite Instability-high) or dMMR (Mismatch Repair Deficient) that might work best to treat these specific cancer types and to understand how well HRO761 is able to treat those cancers.

DETAILED DESCRIPTION:
The new drug being tested in the study, HRO761, is an oral drug that acts on a protein called Werner (WRN), which may contribute to cancer growth. By acting on WRN, HRO761 may be able to stop the growth of the cancer.

This is the first time HRO761 is given to patients and the first time HRO761 is used in combination with pembrolizumab or irinotecan.

Pembrolizumab and irinotecan are drugs approved in several countries and used as standard treatment for certain types of cancer (e.g., colon cancer and small cell lung cancer).

This research study will consist of various treatment arms to investigate HRO761 as single agent and in the combinations.

For HRO761 single agent, the research will be done in two parts. The first part is called "dose escalation" and the second part is called "dose optimization". In the dose escalation part, different groups of people will be given different doses of HRO761 to understand how the body reacts to different doses of the drug and how well the drug acts against the cancer. During the dose optimization part, the selected doses will be tested in more patients until a recommended dose(s) is found.

The combinations of HRO761 with pembrolizumab or irinotecan also will be tested in a dose escalation part to find the recommended doses of HRO761 in these combinations.

Once the recommended doses are determined, more people may be treated with HRO761 alone or together with pembrolizumab or irinotecan to further assess the study treatment effects against various types of MSIhi or dMMR cancers. This part is called dose expansion.

For this research, a number of blood and tissue samples will be collected during the study. Patients may be asked to come approximately 8 times to the clinic during the first 8 weeks and approximately every 2 or 4 weeks thereafter.

Patients will be in the study as long as their study doctor believes that they may be benefiting from the study treatment, unless the patient decides to stop study treatment.

ELIGIBILITY:
Key Inclusion criteria:

* Patients with advanced unresectable or metastatic MSIhi or MMR deficient (dMMR) solid tumors who have progressed after or are intolerant to prior standard therapy.

  * Arm A and C: Patients must have progressed on the most recent therapy for advanced disease including one prior line of immune checkpoint inhibitor therapy.
  * Arm B: Patients should have received prior chemotherapy or targeted therapy, and patients should have received prior immune checkpoint inhibitor or should be expected to benefit from immune checkpoint inhibitor therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Measurable disease as determined by RECIST version 1.1
* • All patients (Arm A, B and C) will have available archival tumor tissue obtained prior to study treatment initiation, to allow retrospective MSIhi/dMMR status confirmation. A newly obtained biopsy will only be collected at screening if there is no archival tumor tissue available and if safe and medically feasible according to treating institution's guidelines. Exceptions may be considered after documented discussion with Novartis.

Key Exclusion criteria:

* Impaired cardiac function or clinically significant cardiac disease
* Clinically significant eye impairment
* Patients with a primary Central Nervous System (CNS) tumor or tumor metastatic to the CNS
* Human Immunodeficiency Virus (HIV) infection
* Active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Tuberculosis infection. Patients whose disease is controlled under antiviral therapy should not be excluded.
* History of severe hypersensitivity reactions to any ingredient of study drug(s)
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., severe ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection), except for prior gastrectomy.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | at month 36
  Month 36 is assumed to be study end.
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Incidence of dose limiting toxicities (DLTs) of treatment (Escalation only) | at Day 28
  A DLT is defined as an adverse event or abnormal laboratory value that is not primarily related to disease, disease progression, intercurrent illness/injury, or concomitant medications that occurs within the first 28 days of study treatment and meets a defined criteria.
Frequency of dose interuptions as a measure of tolerability | at month 36
  Month 36 is assumed to be study end
  Number of dose interruptions by treatment group/arm as a measure of tolerability.
Frequency of dose discontinuations as a measure of tolerability | at month 36
  Month 36 is assumed to be study end
  Number of dose discontinuations by treatment group/arm as a measure of tolerability.
Frequency of dose reductions as a measure of tolerability | at month 36
  Month 36 is assumed to be study end
  Number of dose reductions by treatment group/arm as a measure of tolerability.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per RECIST v1.1 | at month 36
  Month 36 is assumed to be study end
  ORR is the percentage of patients with a best overall response of Complete Response (CR) or Partial Response (PR).
Disease Control Rate (DCR) per RECIST v1.1 | at month 36
  Month 36 is assumed to be study end
  DCR is the percentage of patients with a best overall response of CR or PR or Stable Disease (SD)
Progression Free Survival (PFS) per RECIST v1.1 | at month 36
  Month 36 is assumed to be study end
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause.
Duration of Response (DOR) per RECIST v1.1 | at month 36
  Month 36 is assumed to be study end
  DOR is the time between the date of first documented response (CR or PR) and the date of progression or death due to any cause.
Plasma concentrations of HRO761 | at Day 1, Day 8, Day 29, Day 57, Day 85, Day 113, Day 141, Day 225, and Day 309
  Plasma concentrations of HRO761 will be measured using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) assay.
PK parameter (Tmax) of HRO761 | at month 12
  Cycle 12 (the duration of 1 cycle is 28 days).
  Time to maximum observed concentration (Tmax) determined by non-compartmental PK analysis of plasma concentration-time profiles HRO761.
PK parameter (Cmax) of HRO761 | at month 12
  Cycle 12 (the duration of 1 cycle is 28 days).
  Maximum observed concentration (Cmax) determined by non-compartmental pharmacokinetic (PK) analysis of plasma concentration-time profiles HRO761.
PK parameter (AUC) of HRO761 | at month 12
  Cycle 12 (the duration of 1 cycle is 28 days).
  Area under the plasma concentration-time curve (AUC) determined by non-compartmental PK analysis of plasma concentration-time profiles HRO761.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (6):
  - University of California LA, Los Angeles, California
  - UCSF, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Columbia University Medical Ctr, New York, New York
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Brussels, Belgium
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: No